CLINICAL TRIAL: NCT05091541
Title: A Multicenter Phase I/II Clinical Study on Fully Human Anti-CD19/CD22 Dual Target Chimeric Antigen Receptor Autologous T Cell Injection (CT120) for the Treatment of Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma
Brief Title: A Phase 1/2 Study of CT120 in Patient With Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanjing IASO Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT120C001
Record Dates: First submitted 2021-09-15; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: B-cell Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT120 in relapsed/refractory B-cell non-Hodgkin's lymphoma patients (Experimental): Fully Human Anti-CD19/CD22 Dual Target Chimeric Antigen Receptor Autologous T Cell Injection（CT120）will be infused at 1.0 x 10^6 CAR+ T cells/kg、3.0 x 10^6 CAR+ T cells/kg、6.0 x 10^6 CAR+ T cells/kg in relapsed/refractory B-cell non-Hodgkin's lymphoma patients
  Interventions: Drug: Fully Human Anti-CD19/CD22 Dual Target Chimeric Antigen Receptor Autologous T Cell Injection

INTERVENTIONS:
Drug: Fully Human Anti-CD19/CD22 Dual Target Chimeric Antigen Receptor Autologous T Cell Injection — CT120 is an autologous CD19/22 targeted CAR-T cells injection. The dosage form is a cryopreserved injection solution. The T cells aphesis from subjects then been manufactured to express CAR to binding CD19 and CD22 on B-cell lymphoma.
  Other Names: CT120

SUMMARY:
This study is a single-armed, open-label,multicenter Phase 1/2 study to evaluate the safety and efficacy of CT120 in subjects with relapsed/refractory B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
Leukapheresis procedure will be performed to manufacture CT120. Bridging therapy is allowed between PBMC collection and lymphodepletion. Lymphodepletion with fludarabine and cyclophosphamide was performed for three consecutive days. After 1-day rest, subjects will receive a single dose infusion of CT120. Subjects will be followed in the study for a minimum of 2 years after CT120 infusion. Long-term follow-up for lentiviral vector safety will be followed for up to 15 years after CT120 infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years old.
2. Pathologically confirmed B-cell non-Hodgkin's lymphoma, including:

(1) Diffuse large B-cell lymphoma (DLBCL); (2) Histopathological Grade 3b follicular lymphoma (FL3b); (3) Follicular lymphoma with diffuse large B cell transformation; (4) Primary mediastinal large B-cell lymphoma (PMBCL). 3. Relapsed/refractory B-cell non-Hodgkin's lymphoma must meet one of the following criteria:

1. At least 2 failed prior B-cell non-Hodgkin's lymphoma treatment regimens (including relapse, no response, and progression). Prior therapy must have included anti-CD20 monoclonal antibodies (except for CD20-negative subjects) and standard therapies which including anthracyclines;
2. Recurrence after autologous hematopoietic stem cell transplantation;
3. Primary resistance: After 2 cycles of initial anti-CD20 monoclonal immunochemotherapy, the best response was stable disease or disease progression.

4. At least 1 measurable lesion as following:

1. The long axis of the lymph node lesions should be ≥15mm (and the length of the short axis is measurable), or;
2. The lengths of extra-lymph node lesions should be ≥10mm in both the long and short axis.

5. Expected survival time≥12 weeks. 6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. 7. Adequate organ function before enrollment, and meet all the following laboratory test results:

1. Blood routine: neutrophils ≥1.0 ×109/L (granulocyte colony stimulating factor (G-CSF) is allowed within 7 days before the examination), lymphocytes ≥0.3 ×109 /L, platelets ≥50 ×109 /L (must have not received blood transfusion [including component transfusion] or treatments that include thrombopoietin [TPO] for the purpose of raising platelets within 7 days before the examination), hemoglobin ≥80g/L (must have not received blood transfusion [including component blood transfusion] within 7 days before the examination);
2. Blood coagulation function: fibrinogen≥1.0g/L; activated partial thromboplastin time≤1.5×ULN, prothrombin time (PT)≤1.5×ULN;
3. Liver function: ALT and AST≤2.5×ULN; serum total bilirubin≤1.5×ULN;
4. Renal function: creatinine clearance rate CrCl ≥60 mL/min estimated by Cockcroft-Gault;
5. Left ventricular ejection fraction (LVEF)≥50% estimated by echocardiography;
6. Baseline oxygen saturation > 91% on room air. 8. Females and males with childbearing potential should take effective contraception from the day of signing the informed consent form to 365 days after the CT120 infusion. Effective contraception is defined as: abstinence or contraceptive methods with an annual failure rate of <1% indicated in section 9.8 of this protocol.

9. Subject is willing to participate in this trial and sign an informed consent form.

Exclusion Criteria:

1. Subjects who have received or require the following treatments:

(1) Prior CAR-T cell therapy before enrollment; (2) Presence of acute or chronic graft-versus-host disease (GVHD) requires systemic treatment within 4 weeks before enrollment; (3) History of immunodeficiency or other diseases and autoimmune diseases (eg Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus, etc.) received immunosuppressive therapy within 2 years before enrollment; (4) Autologous hematopoietic stem cell transplantation (autoSCT) within 12 weeks before enrollment and history of allogeneic stem cell transplantation (HSCT); (5) Live vaccines injection within 4 weeks before enrollment; (6) According to investigator's discretion, there is a need to use systemic corticosteroid therapy within 12 weeks after the administration of the study drug (except for hydrocortisone ≤12mg/m2/day or other hormones converting into the same dose range for physiological replacement therapy) or other immunosuppressive drug therapy (except local therapy).

2. B-cell non-Hodgkin's lymphoma patients with active central nervous system or intestinal parenchyma invasion.

3. Excessive tumor burden and any lesions with a long axis ≥10cm. 4. Other active malignant tumors in the past 5 years, except for curable tumor that has been completely cured, such as basal or squamous cell carcinoma, cervical or breast carcinoma in situ, etc.

5. Positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and an abnormal HBV DNA result detected by peripheral blood test (abnormal HBV DNA result is defined as: the quantitative detection of HBV DNA is over the detectable lower limit or beyond the normal reference of the testing center or HBV viral DNA positive); Hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA positive; Human immunodeficiency virus (HIV) antibody positive; Cytomegalovirus (CMV) DNA test positive; syphilis test positive.

6. Uncontrollable active infections (except for genitourinary system infections and upper respiratory tract infections < CTCAE Grade 2).

7. Severe heart disease: including but not limited to unstable angina, myocardial infarction (within 6 months before screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ Grade III), severe arrhythmia.

8. Hypertension that cannot be controlled by medication. 9. Adverse events during prior therapies have not relieved to baseline or ≤1 (according to NCI-CTCAE v5.0, except for alopecia).

10. Major surgery within 2 weeks before enrollment, or surgeries that were planed while waiting for infusion or within 12 weeks after receiving investigational product (except planned local anesthesia surgery).

11. History of organ transplant. 12. Pregnant or lactating women. 13. Previous central nervous system diseases (such as cerebral aneurysm, epilepsy, stroke, Alzheimer's disease, mental illness, etc.) or mental disorders.

14. Unstable systemic diseases judged by other researchers: including but not limited to severe liver, kidney, or metabolic diseases that require medication.

15. Other unsuitable situations for enrollment judged by investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2021-10-20 (Estimated); Primary Completion 2024-10-20 (Estimated); Study Completion 2039-10-20 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Types and incidence of Dose-limiting toxicity (DLT) | up to 28 days after CT120 infusion
  Dose-limiting toxicity (DLT) will be collected and graded according to American Society for Transplantation and Cellular Therapy (ASTCT) consensus (for CRS/ICANS) and CTCAE v5.0(for AE except CRS/ICANS)
Phase 1:Types and incidence of adverse events (AEs) ，serious adverse events (SAEs) and adverse events of special interest (AESI) | Up to 2 years after CT120 CAR T-cells infusion
  AE will be collected and graded according to American Society for Transplantation and Cellular Therapy (ASTCT) consensus (for CRS/ICANS) and CTCAE v5.0(for AE except CRS/ICANS)
Phase 2:Overall response rate (ORR) at Day 90 | Up to 90 Days after CT120 infusion
  ORR will be calculated as the percentage of patients who achieved partial response (PR) or better at Day 90

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to Day 28、Day 90、Day180 after CT120 infusion
  ORR will be calculated as the percentage of patients who achieved partial response (PR) or better.
Time to Response (TTR) | Up to 2 years after CT120 infusion
  Time from CT120 infusion to first documentation of response.
Time to complete Response (TTCR) | Up to 2 years after CT120 infusion
  Time from CT120 infusion to first documentation of complete response.
Duration of Response (DOR) | Up to 2 years after CT120 infusion
  Time from first response to disease progression or death from any cause
Progression-free Survival (PFS) | Up to 2 years after CT120 infusion
  PFS will be calculated as the time from CT120 infusion to disease progression or death from any cause (whichever occurs first).
Overall Survival (OS) | Up to 2 years after CT120 infusion
  Time from CT120 infusion to time of death due to any cause
Quantity of CAR copies in peripheral blood | Up to 2 years after CT120 infusion
  CAR copies in peripheral blood will be measured by quantitative polymerase chain reaction (qPCR) in 2 years.
Quantity of CAR T-cells level in peripheral blood | Up to 2 years after CT120 infusion
  CAR T-cells in peripheral blood will be measured by flow cytometry (FCM) in 2 years
Laboratory tests | Up to 2 years after CT120 infusion
  Abnormal results of laboratory tests
Vital signs | Up to 2 years after CT120 infusion
  Abnormal results of vital signs
Physical examination | Up to 2 years after CT120 infusion
  Abnormal results of physical examination

OTHER OUTCOMES:
Immunogenicity | Up to 2 years after CT120 infusion
  Development of an anti-CAR antibody response
Replication competent lentivirus (RCL) | Up to 15 years after CT120 infusion
  The incidence of replication competent lentivirus (RCL)
Changes in the proportion of peripheral blood lymphocyte subsets | Up to 2 years after CT120 infusion
  Changes in the proportion of lymphocyte subsets in the peripheral blood will be analyzed by immune cell phenotyping using flow cytometry.
Correlation between cytokines/inflammation-related proteins and Incidence of Adverse Event | Up to 2 years after CT120 infusion
Correlation between cytokines/inflammation-related proteins and efficacy | Up to 2 years after CT120 infusion
Correlation between efficacy and CD19/CD22 antigen expression in tumor tissues | Up to 2 years after CT120 infusion
Correlation between efficacy and gene mutations including MYC, BCL2 and BCL6 rearrangements | Up to 2 years after CT120 infusion
Correlation between efficacy and and the expression of oncogenes including C-myc and BCL | Up to 2 years after CT120 infusion